CLINICAL TRIAL: NCT03649594
Title: Risk Stratification for Subclinical Leaflet Thrombosis Post TAVI Using Thromboelastography
Brief Title: Risk Stratification Post TAVI Using TEG
Acronym: RISTRATAVI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Torben Pottgiesser (Other)
Responsible Party: Sponsor-Investigator, Torben Pottgiesser, PD Dr. (Assistant Professor), University Hospital Freiburg
Organization: University Hospital Freiburg (Other)
Other Study IDs: RISTRATAVI-1-2019
Record Dates: First submitted 2018-08-10; First posted 2018-08-28 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Platelet Function Tests; Predictive Value of Tests; Thrombelastography; Cardiovascular Diseases; Aortic Valve Stenosis; Thrombosis; Transcatheter Aortic Valve Replacement
MeSH Terms: conditions — Cardiovascular Diseases; Aortic Valve Stenosis; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- TAVI and no therapeutic anticoagulation: Subjects in this group do not have an indication for therapeutic anticoagulation.
- TAVI and therapeutic anticoagulation: Subjects in this group have an indication for therapeutic anticoagulation such as atrial fibrillation.

SUMMARY:
Transcatheter aortic valve implantation (TAVI) has become the standard of care in elderly patients at increased risk for surgical aortic valve replacement . However, the optimal antithrombotic strategy post TAVI is still unclear. Current European guidelines recommend dual antiplatelet therapy (DAPT) for 3 to 6 months.The prevalence of subclinical leaflet thrombosis after TAVI is 15% up to 40%, but its clinical long-term relevance is uncertain. Thromboelastography (TEG(R)) can be used as a point-of-care system evaluating a patient's individual hemostasis profile. For the detection of transcatheter valve thrombosis it may be superior to conventional platelet function testing because global hemostasis can be assessed in addition to platelet function. The investigators intend an observational trial recruiting patients undergoing TAVI under standard care. At defined time points the investigators will serially perform TEG(R) as well as further platelet function testing (multiple electrode aggregometry) and conventional coagulation testing. The primary objective is to find surrogate TEG-derived markers / models predicting the development of a subclinical leaflet thrombosis after TAVI under usual care. The secondary objective is to find TEG-derived markers / models identifying patients at an increased risk after TAVI (all-cause mortality, cardiovascular mortality, thromboembolic and bleeding events).

DETAILED DESCRIPTION:
Aortic stenosis is the most common primary valve disease in high-income countries with increasing importance. Throughout the last 15 years, transcatheter aortic valve implantation (TAVI) has become an alternative to surgical aortic valve replacement, the former standard of care. Nowadays, the use of TAVI in elderly patients at increased surgical risk is favored. There is still an important lack of evidence concerning the optimal antithrombotic strategy post TAVI. Recently, it has been shown that the prevalence of subclinical leaflet thrombosis after intervention has been underestimated and may be present in around 15 % up to 40% (PORTICO IDE trial) of transcatheter valves. One study demonstrated that transient ischemic attacks are significantly increased in these patients.

European guidelines are undecided towards the length of the dual antiplatelet therapy (DAPT) after TAVI and recommend optional treatment durations between 3 to 6 months. The optimal duration of DAPT is not known, although DAPT duration is associated with an increased bleeding risk. The most recent update of AHA guidelines for valvular heart disease state that oral anticoagulation with a VKA (INR of 2.5) may be reasonable for at least 3 months after TAVI in patients at low risk of bleeding. Without favoring one over the other recommendation, the current AHA guidelines also maintain the prior statement (from 2014) that clopidogrel 75 mg daily may be reasonable for the first 6 months after TAVI in addition to life-long aspirin, which is in accordance with the European Guideline recommendation. On the other hand, the GALILEO trial has recently been stopped as patients receiving rivaroxaban after TAVI (no prior atrial fibrillation) had a higher mortality and thromboembolic events as well as higher bleeding event rates.

The TEG(R) 6S analyzer is a point-of-care system evaluating a patient's individual hemostasis profile by thrombelastography (TEG(R)), a potentially superior tool compared to conventional platelet function testing. The TEG(R) system has been able to predict thrombotic complications in different clinical contexts.

In classic coronary interventional cardiology, the strength of adenosine diphosphate (ADP)-induced and thrombin-induced platelet-fibrin clots were found to be indicators of long-term poststenting ischemic events. As the pathophysiologic mechanism of subclinical leaflet thrombosis has not been examined in detail, the investigators hypothesize that several TEG(R) assays may provide insight in finding predictive TEG(R) markers. Furthermore, as the onset of subclinical leaflet thrombosis is not clear and may possibly increase over time, the design with subsequent TEG(R) analyses at 3 timepoints (0, 3, 6 months) will help to hopefully identify predictors that may become evident at later time points.

It is intriguing to hypothesize that the better predictive marker may be found using the Global Hemostasis Assay. This is relevant as leaflet thrombosis develops despite dual antiplatelet therapy and anticoagulation has been shown to fully resolve subclinical leaflet thrombosis. The Global Hemostasis Assay may deliver prediction beyond platelet function, which may improve antithrombotic therapy post TAVI. Finding a predictive TEG marker (examining Platelet Mapping and Global Hemostasis together) holds the promise for future individualized clinical decision-making by identifying individual risk.

Taken together, we hope that individual TEG based stratification of patients at risk for subclinical leaflet thrombosis or other events may allow individual clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

- Patients are eligible for enrollment if they are scheduled for TAVI using a commercially available valve after clinical decision making within the local Heart Team.

Exclusion Criteria:

* Valve-in-valve TAVI and prior valve thrombosis
* Severely impaired renal function (e.g. creatinine clearance < 30ml/min)
* poor CT imaging if the presence of HALT cannot be assessed.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that are scheduled for TAVI using a commercially available valve after clinical decision making within the local Heart Team will be possible subjects yielding the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Global TEG(R)-based prediction of hypoattenuating leaflet thickening (HALT) | 6 months
  TEG(R)readout Global Hemostasis Assay
Platelet TEG(R)-based prediction of hypoattenuating leaflet thickening (HALT) | 6 months
  TEG(R)readout Platelet Mapping Assay

SECONDARY OUTCOMES:
All-cause mortality within 12 months | 12 months
  All-cause mortality will be recorded within 12 months after TAVI.
Cardiovascular mortality within 12 months | 12 months
  Cardiovascular mortality will be recorded within 12 months after TAVI.
Thromboembolic events within 12 months | 12 months
  Thromboembolic events will be recorded within 12 months after TAVI.
Bleeding events within 12 months | 12 months
  Bleeding events will be recorded within 12 months after TAVI.

OTHER OUTCOMES:
Incidence of hypoattenuating leaflet thickening (HALT) | 6 months
  Presence of HALT on CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Torben Pottgiesser, MD, Principal Investigator — Cardiology and Angiology I, Heart Center Freiburg University, Germany; Daniel Duerschmied, MD, Study Director — Cardiology and Angiology I, Heart Center Freiburg University, Germany
Locations (1):
- Department of Cardiology and Angiology I, Heart Center Freiburg University, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ben-Dor I, Pichard AD, Gonzalez MA, Weissman G, Li Y, Goldstein SA, Okubagzi P, Syed AI, Maluenda G, Collins SD, Delhaye C, Wakabayashi K, Gaglia MA Jr, Torguson R, Xue Z, Satler LF, Suddath WO, Kent KM, Lindsay J, Waksman R. Correlates and causes of death in patients with severe symptomatic aortic stenosis who are not eligible to participate in a clinical trial of transcatheter aortic valve implantation. Circulation. 2010 Sep 14;122(11 Suppl):S37-42. doi: 10.1161/CIRCULATIONAHA.109.926873. PMID 20837923
- [Background] Hamm CW, Arsalan M, Mack MJ. The future of transcatheter aortic valve implantation. Eur Heart J. 2016 Mar 7;37(10):803-10. doi: 10.1093/eurheartj/ehv574. Epub 2015 Nov 17. PMID 26578195
- [Background] Ruile P, Jander N, Blanke P, Schoechlin S, Reinohl J, Gick M, Rothe J, Langer M, Leipsic J, Buettner HJ, Neumann FJ, Pache G. Course of early subclinical leaflet thrombosis after transcatheter aortic valve implantation with or without oral anticoagulation. Clin Res Cardiol. 2017 Feb;106(2):85-95. doi: 10.1007/s00392-016-1052-3. Epub 2016 Nov 16. PMID 27853942
- [Background] Yanagisawa R, Hayashida K, Yamada Y, Tanaka M, Yashima F, Inohara T, Arai T, Kawakami T, Maekawa Y, Tsuruta H, Itabashi Y, Murata M, Sano M, Okamoto K, Yoshitake A, Shimizu H, Jinzaki M, Fukuda K. Incidence, Predictors, and Mid-Term Outcomes of Possible Leaflet Thrombosis After TAVR. JACC Cardiovasc Imaging. 2016 Dec 8:S1936-878X(16)30897-X. doi: 10.1016/j.jcmg.2016.11.005. Online ahead of print. PMID 28017712
- [Background] Makkar RR, Fontana G, Jilaihawi H, Chakravarty T, Kofoed KF, De Backer O, Asch FM, Ruiz CE, Olsen NT, Trento A, Friedman J, Berman D, Cheng W, Kashif M, Jelnin V, Kliger CA, Guo H, Pichard AD, Weissman NJ, Kapadia S, Manasse E, Bhatt DL, Leon MB, Sondergaard L. Possible Subclinical Leaflet Thrombosis in Bioprosthetic Aortic Valves. N Engl J Med. 2015 Nov 19;373(21):2015-24. doi: 10.1056/NEJMoa1509233. Epub 2015 Oct 5. PMID 26436963
- [Background] Chakravarty T, Sondergaard L, Friedman J, De Backer O, Berman D, Kofoed KF, Jilaihawi H, Shiota T, Abramowitz Y, Jorgensen TH, Rami T, Israr S, Fontana G, de Knegt M, Fuchs A, Lyden P, Trento A, Bhatt DL, Leon MB, Makkar RR; RESOLVE; SAVORY Investigators. Subclinical leaflet thrombosis in surgical and transcatheter bioprosthetic aortic valves: an observational study. Lancet. 2017 Jun 17;389(10087):2383-2392. doi: 10.1016/S0140-6736(17)30757-2. Epub 2017 Mar 19. PMID 28330690
- [Background] Baumgartner H, Falk V, Bax JJ, De Bonis M, Hamm C, Holm PJ, Iung B, Lancellotti P, Lansac E, Rodriguez Munoz D, Rosenhek R, Sjogren J, Tornos Mas P, Vahanian A, Walther T, Wendler O, Windecker S, Zamorano JL; ESC Scientific Document Group. 2017 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2017 Sep 21;38(36):2739-2791. doi: 10.1093/eurheartj/ehx391. No abstract available. PMID 28886619
- [Background] Valgimigli M, Campo G, Monti M, Vranckx P, Percoco G, Tumscitz C, Castriota F, Colombo F, Tebaldi M, Fuca G, Kubbajeh M, Cangiano E, Minarelli M, Scalone A, Cavazza C, Frangione A, Borghesi M, Marchesini J, Parrinello G, Ferrari R; Prolonging Dual Antiplatelet Treatment After Grading Stent-Induced Intimal Hyperplasia Study (PRODIGY) Investigators. Short- versus long-term duration of dual-antiplatelet therapy after coronary stenting: a randomized multicenter trial. Circulation. 2012 Apr 24;125(16):2015-26. doi: 10.1161/CIRCULATIONAHA.111.071589. Epub 2012 Mar 21. PMID 22438530
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Fleisher LA, Jneid H, Mack MJ, McLeod CJ, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A. 2017 AHA/ACC Focused Update of the 2014 AHA/ACC Guideline for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2017 Jul 11;70(2):252-289. doi: 10.1016/j.jacc.2017.03.011. Epub 2017 Mar 15. No abstract available. PMID 28315732
- [Background] Parker RJ, Eley KA, Von Kier S, Pearson O, Watt-Smith SR. Functional fibrinogen to platelet ratio using thromboelastography as a predictive parameter for thrombotic complications following free tissue transfer surgery: a preliminary study. Microsurgery. 2012 Oct;32(7):512-9. doi: 10.1002/micr.21978. Epub 2012 Mar 31. PMID 22473821
- [Background] Krzanicki D, Sugavanam A, Mallett S. Intraoperative hypercoagulability during liver transplantation as demonstrated by thromboelastography. Liver Transpl. 2013 Aug;19(8):852-61. doi: 10.1002/lt.23668. Epub 2013 Jul 8. PMID 23696318
- [Background] Gurbel PA, Bliden KP, Navickas IA, Mahla E, Dichiara J, Suarez TA, Antonino MJ, Tantry US, Cohen E. Adenosine diphosphate-induced platelet-fibrin clot strength: a new thrombelastographic indicator of long-term poststenting ischemic events. Am Heart J. 2010 Aug;160(2):346-54. doi: 10.1016/j.ahj.2010.05.034. PMID 20691842
- [Background] Pache G, Schoechlin S, Blanke P, Dorfs S, Jander N, Arepalli CD, Gick M, Buettner HJ, Leipsic J, Langer M, Neumann FJ, Ruile P. Early hypo-attenuated leaflet thickening in balloon-expandable transcatheter aortic heart valves. Eur Heart J. 2016 Jul 21;37(28):2263-71. doi: 10.1093/eurheartj/ehv526. Epub 2015 Oct 7. PMID 26446193
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343